CLINICAL TRIAL: NCT02586805
Title: HELP Study: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Efficacy and Safety Study to Evaluate DX-2930 For Long-Term Prophylaxis Against Acute Attacks of Hereditary Angioedema (HAE)
Brief Title: Efficacy and Safety Study of DX-2930 to Prevent Acute Angioedema Attacks in Patients With Type I and Type II HAE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Collaborators: Dyax Corp. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DX-2930-03; 2015-003943-20 (EudraCT Number)
Record Dates: First submitted 2015-10-23; First posted 2015-10-26 (Estimated); Results first posted 2018-04-24 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Hereditary Angioedema (HAE)
Keywords: DX-2930; Hereditary Angioedema; Dyax
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — lanadelumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- DX-2930 300 mg every 2 weeks (Experimental): 300 mg DX-2930 administered every 2 weeks by subcutaneous injection.
  Interventions: Drug: DX-2930 - 300mg/2wk
- DX-2930 300 mg every 4 weeks (Experimental): 300 mg DX-2930 administered every 4 weeks by subcutaneous injection
  Interventions: Drug: DX-2930 - 300mg/4wk
- DX-2930 150 mg every 4 weeks (Experimental): 150 mg DX-2930 administered every 4 weeks by subcutaneous injection
  Interventions: Drug: DX-2930 - 150mg/4wk
- Placebo (Placebo Comparator): Placebo administered every 2 weeks by subcutaneous injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DX-2930 - 300mg/2wk — 300 mg DX-2930 administered every 2 weeks by subcutaneous injection.
  Arms: DX-2930 300 mg every 2 weeks
Drug: DX-2930 - 300mg/4wk — 300 mg DX-2930 administered every 4 weeks by subcutaneous injection. To maintain the study blind, subjects will be given placebo injections every other 2 weeks when they are not receiving drug.
  Arms: DX-2930 300 mg every 4 weeks
Drug: DX-2930 - 150mg/4wk — 150 mg DX-2930 administered every 4 weeks by subcutaneous injection. To maintain the study blind, subjects will be given placebo injections every other 2 weeks when they are not receiving drug.
  Arms: DX-2930 150 mg every 4 weeks
Drug: Placebo — Placebo administered every 2 weeks by subcutaneous injection.
  Arms: Placebo

SUMMARY:
This is a phase 3, multicenter, randomized, double-blind, placebo-controlled trial to evaluate the efficacy and safety of DX-2930 in preventing acute angioedema attacks in patients with Type I and Type II HAE.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 12 years of age or older at time of screening
* Documented diagnosis of HAE, Type I or II
* Baseline rate of at least 1 Investigator-confirmed HAE attack per 4 weeks
* Adult subjects and caregivers of subjects under the age of 18 are willing and able to read, understand, and sign an informed consent form. Subjects age 12 to 17, whose caregiver provides informed consent, are willing and able to read, understand an dsign an assent form.
* Males and femailes who are fertile and sexually active must adhere to contraception requirements.

Exclusion Criteria:

* Concomitant diagnosis of another form of chronic, recurrent angioedema, such as acquired angioedema, idiopathic angioedema, or recurrent angioedema associated with urticaria.
* Participation in a prior DX-2930 study
* Treatment with any other investigational drug or exposure to an investigational device within 4 weeks prior screening
* Exposure to angiotensin-converting enzyme (ACE) inhibitors or any estrogen-containing medications within 4 weeks prior to screening.
* Exposure to androgens within 2 weeks prior to entering the run-in period.
* Use of long-term prophylactic therapy for HAE within 2 weeks prior to entering the run-in period.
* Use of short-term prophylaxis for HAE within 7 days prior to entering the run-in period.
* Any of the following liver function test abnormalities: alanine aminotransferase (ALT) > 3x upper limit of normal, or aspartate aminotransferase (AST) > 3x upper limit of normal, or total bilirubin > 2x upper limit of normal (unless the bilirubin elevation is a result of Gilbert's syndrome).
* Pregnancy or breastfeeding.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2017-04-13 (Actual); Study Completion 2017-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shire Physician, Study Director — Shire
Locations (41):
- United States (31):
  - Clinical Research Center of Alabama, LLC, Birmingham, Alabama
  - Medical Research of Arizona, Scottsdale, Arizona
  - UC San Diego School of Medicine, San Diego, California
  - AIRE Medical of Los Angeles, Santa Monica, California
  - Allergy & Asthma Clinical Research, Walnut Creek, California
  - IMMUNOe International Health & Research Centers, Centennial, Colorado
  - Asthma and Allergy Associates, P.C., Colorado Springs, Colorado
  - University of South Florida, Tampa, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Institute of Asthma & Allergy, P.C., Chevy Chase, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Hospital and Health System, Ann Arbor, Michigan
  - Midwest Immunology Clinic, Plymouth, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hudson-Essex Allergy, LLC, Belleville, New Jersey
  - Atlantic Research Center, LLC, Ocean City, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - The Mount Sinai Medical Center, New York, New York
  - American Health Research, Charlotte, North Carolina
  - Duke Asthma, Allergy and Airway Center, Durham, North Carolina
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Optimed Research, LTD, Columbus, Ohio
  - Toledo Institute of Clinical Research, Toledo, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Austin Regional Clinic, Austin, Texas
  - AARA Research Center, Dallas, Texas
  - Intermountain Clinical Research, Draper, Utah
  - Allergy Associates of Utah, Murray, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Marycliff Allergy Specialists, Spokane, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - Ottawa Allergy Research Corporation, Ottawa, Ontario
  - Gordon Sussman Clinical Research Inc., Toronto, Ontario
  - Clinique Specialisee en Allergie de la Capitale, Québec, Quebec
- Germany (3):
  - Charité - University of Berlin, Berlin
  - Hautklinik und Poliklinik der Universitätsmedizin, Mainz
  - HZRM Hamophilie-Zentrum Rhein Main, Mörfelden-Walldorf
- Hospital L. Sacco, Milan University, Milan, Italy
- Triumpharma, Amman, Jordan
- Sociedad Alergologica, San Juan, PR, Puerto Rico
- Barts Health NHS Trust Clinical Research Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Lumry WR, Maurer M, Weller K, Riedl MA, Watt M, Yu M, Devercelli G, Meunier J, Banerji A; HELP OLE Study Group. Long-term lanadelumab treatment improves health-related quality of life in patients with hereditary angioedema. Ann Allergy Asthma Immunol. 2023 Jul;131(1):101-108.e3. doi: 10.1016/j.anai.2023.03.028. Epub 2023 Apr 5. PMID 37028510
- [Derived] Beard N, Frese M, Smertina E, Mere P, Katelaris C, Mills K. Interventions for the long-term prevention of hereditary angioedema attacks. Cochrane Database Syst Rev. 2022 Nov 3;11(11):CD013403. doi: 10.1002/14651858.CD013403.pub2. PMID 36326435
- [Derived] Craig TJ, Zaragoza-Urdaz RH, Li HH, Yu M, Ren H, Juethner S, Anderson J; HELP and HELP OLE Study Investigators. Effectiveness and safety of lanadelumab in ethnic and racial minority subgroups of patients with hereditary angioedema: results from phase 3 studies. Allergy Asthma Clin Immunol. 2022 Sep 24;18(1):85. doi: 10.1186/s13223-022-00721-y. PMID 36153561
- [Derived] Banerji A, Riedl MA, Bernstein JA, Cicardi M, Longhurst HJ, Zuraw BL, Busse PJ, Anderson J, Magerl M, Martinez-Saguer I, Davis-Lorton M, Zanichelli A, Li HH, Craig T, Jacobs J, Johnston DT, Shapiro R, Yang WH, Lumry WR, Manning ME, Schwartz LB, Shennak M, Soteres D, Zaragoza-Urdaz RH, Gierer S, Smith AM, Tachdjian R, Wedner HJ, Hebert J, Rehman SM, Staubach P, Schranz J, Baptista J, Nothaft W, Maurer M; HELP Investigators. Effect of Lanadelumab Compared With Placebo on Prevention of Hereditary Angioedema Attacks: A Randomized Clinical Trial. JAMA. 2018 Nov 27;320(20):2108-2121. doi: 10.1001/jama.2018.16773. PMID 30480729

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 41 sites in the United States, United Kingdom, Italy, Germany, Canada and Jordan between 03 March 2016 (first participant first visit) and 13 April 2017 (last participant last visit).
Pre-assignment Details: A total of 159 participants were screened and 126 participants were randomized in the ratio of 3:2:2:2 to the placebo versus DX-2930-03 arms. Of them, 125 participants were assigned to study treatment and one participant determined to be screen failure after randomization.
Groups:
- Placebo: Participants received placebo matched to DX-2930 subcutaneously (SC) once in every 2 weeks (q2wks) for 26 weeks.
- Lanadelumab (DX-2930) 150 mg Every 4 Weeks: Participants received 150 milligram (mg) dose of DX-2930 SC once in every 4 weeks (q4wks) and matched placebo SC q2wks between DX-2930 doses for 26 weeks.
- Lanadelumab (DX-2930) 300 mg Every 4 Weeks: Participants received 300 mg dose of DX-2930 SC q4wks and matched placebo SC q2wks between DX-2930 doses for 26 weeks.
- Lanadelumab (DX-2930) 300 mg Every 2 Weeks: Participants received 300 mg dose of DX-2930 SC q2wks for 26 weeks.
Period: Overall Study
Arm/Group | Placebo | Lanadelumab (DX-2930) 150 mg Every 4 Weeks | Lanadelumab (DX-2930) 300 mg Every 4 Weeks | Lanadelumab (DX-2930) 300 mg Every 2 Weeks
Started | 41 | 28 | 29 | 27
Completed | 35 | 27 | 26 | 25
Not Completed | 6 | 1 | 3 | 2
Not completed — Withdrawal by Subject | 3 | 1 | 1 | 2
Not completed — Adverse Event | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants who received any exposure to the investigational product.
Groups:
- Placebo: Participants received placebo matched to DX-2930 SC q2wks for 26 weeks.
- Lanadelumab (DX-2930) 150 mg Every 4 Weeks: Participants received 150 mg dose of DX-2930 SC q4wks and matched placebo SC q2wks between DX-2930 doses for 26 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Lanadelumab (DX-2930) 150 mg Every 4 Weeks | Lanadelumab (DX-2930) 300 mg Every 4 Weeks | Lanadelumab (DX-2930) 300 mg Every 2 Weeks | Total
Number analyzed (Participants) | 41 | 28 | 29 | 27 | 125
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.1 (16.75) | 43.4 (14.91) | 39.5 (12.85) | 40.3 (13.35) | 40.7 (14.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 20 | 19 | 15 | 88
  Male | 7 | 8 | 10 | 12 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 2 | 3 | 9
  Not Hispanic or Latino | 38 | 27 | 27 | 23 | 115
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Investigator Confirmed Hereditary Angioedema (HAE) Attacks During Treatment Period
Description: HAE attack was defined as a discrete episode during which the participant progressed from no angioedema to symptoms of angioedema. Rate of investigator confirmed HAE attacks was analyzed using a generalized linear model (GLM) for count data assuming a poisson distribution with a log link function and Pearson chi-square scaling of standard errors to account for potential overdispersion. The logarithm of time in days each subject was observed during the treatment period was used as an offset variable in the model.
Time Frame: From Day 0 to Day 182
Population: ITT population included all randomized participants who received any exposure to the investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: Attacks per 4 weeks
Arm/Group | Placebo | Lanadelumab (DX-2930) 150 mg Every 4 Weeks | Lanadelumab (DX-2930) 300 mg Every 4 Weeks | Lanadelumab (DX-2930) 300 mg Every 2 Weeks
Number analyzed (Participants) | 41 | 28 | 29 | 27
Attacks per 4 weeks | 1.967 [1.640 to 2.358] | 0.480 [0.313 to 0.735] | 0.526 [0.358 to 0.771] | 0.257 [0.145 to 0.458]
Statistical Analysis 1: Comparison: Placebo vs Lanadelumab (DX-2930) 150 mg Every 4 Weeks; Test type: Other; p < 0.001, Chi-squared — p-values are adjusted for multiple testing; % change in mean rate (vs placebo) = -75.609, 95% CI 2-sided [-84.650 to -61.243] — % change in mean rate corresponds to 100% * (estimated mean rate ratio - 1); Results from Poisson regression model with fixed effects for treatment group (categorical) and normalized baseline attack rate (continuous), and logarithm of time in days each participant was observed during treatment period as offset variable in model. Pearson chi-square scaling of standards errors was employed to account for potential overdispersion. Mean estimates are Least Squares (LS) means
Statistical Analysis 2: Comparison: Placebo vs Lanadelumab (DX-2930) 300 mg Every 4 Weeks; Test type: Other; p < 0.001, Chi-squared — p-values are adjusted for multiple testing; % change in mean rate (vs placebo) = -73.271, 95% CI 2-sided [-82.379 to -59.456] — % change in mean rate corresponds to 100% * (estimated mean rate ratio - 1); [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Lanadelumab (DX-2930) 300 mg Every 2 Weeks; Test type: Other; p < 0.001, Chi-squared — p-values are adjusted for multiple testing; % change in mean rate (vs placebo) = -86.921, 95% CI 2-sided [-92.828 to -76.150] — % change in mean rate corresponds to 100% * (estimated mean rate ratio - 1); [other analysis details as in outcome 1, analysis 1]

2. Secondary Outcome: Rate of Investigator Confirmed Hereditary Angioedema (HAE) Attack Requiring Acute Treatment
Description: HAE attack was defined as a discrete episode during which the participant progressed from no angioedema to symptoms of angioedema. Rate of investigator confirmed HAE attack was analyzed using the GLM for count data assuming a poisson distribution with a log link function and Pearson chi-square scaling of standard errors to account for potential overdispersion. The logarithm of time in days each subject was observed during the treatment period was used as an offset variable in the model.
Time Frame: From Day 0 to Day 182
Population: ITT population included all randomized participants who received any exposure to the investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: Attacks per 4 weeks
Arm/Group | Placebo | Lanadelumab (DX-2930) 150 mg Every 4 Weeks | Lanadelumab (DX-2930) 300 mg Every 4 Weeks | Lanadelumab (DX-2930) 300 mg Every 2 Weeks
Number analyzed (Participants) | 41 | 28 | 29 | 27
Attacks per 4 weeks | 1.637 [1.337 to 2.005] | 0.314 [0.184 to 0.535] | 0.423 [0.276 to 0.648] | 0.208 [0.109 to 0.396]
Statistical Analysis 1: Comparison: Placebo vs Lanadelumab (DX-2930) 150 mg Every 4 Weeks; Test type: Other; p < 0.001, Chi-squared — p-values are adjusted for multiple testing; % change in mean rate (vs placebo) = -80.842, 95% CI 2-sided [-89.169 to -66.114] — % change in mean rate corresponds to 100% * (estimated mean rate ratio - 1); [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Lanadelumab (DX-2930) 300 mg Every 4 Weeks; Test type: Other; p < 0.001, Chi-squared — p-values are adjusted for multiple testing; % change in mean rate (vs placebo) = -74.169, 95% CI 2-sided [-83.733 to -58.983] — % change in mean rate corresponds to 100% * (estimated mean rate ratio - 1); [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Lanadelumab (DX-2930) 300 mg Every 2 Weeks; Test type: Other; p < 0.001, Chi-squared — p-values are adjusted for multiple testing; % change in mean rate (vs placebo) = -87.299, 95% CI 2-sided [-93.494 to -75.204] — % change in mean rate corresponds to 100% * (estimated mean rate ratio - 1); [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Rate of Moderate or Severe Investigator Confirmed Hereditary Angioedema (HAE) Attacks
Description: HAE attack was defined as a discrete episode during which the participant progressed from no angioedema to symptoms of angioedema. Moderate and severe investigator-confirmed HAE attacks were the attacks that were moderate or severe as per the HAE attack assessment and reporting procedures (HAARP) defined severity. The overall severity of attack was determined by the investigator using following definitions: mild (transient or mild discomfort), moderate (mild to moderate limitation in activity), severe (marked limitation in activity). Rate of moderate or severe investigator confirmed HAE attack was analyzed using the GLM for count data assuming a poisson distribution with a log link function and Pearson chi-square scaling of standard errors to account for potential overdispersion. The logarithm of time in days each subject was observed during the treatment period was used as an offset variable in the model.
Time Frame: From Day 0 to Day 182
Population: ITT population included all randomized participants who received any exposure to the investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: Attacks per 4 weeks
Arm/Group | Placebo | Lanadelumab (DX-2930) 150 mg Every 4 Weeks | Lanadelumab (DX-2930) 300 mg Every 4 Weeks | Lanadelumab (DX-2930) 300 mg Every 2 Weeks
Number analyzed (Participants) | 41 | 28 | 29 | 27
Attacks per 4 weeks | 1.216 [0.971 to 1.522] | 0.359 [0.221 to 0.581] | 0.325 [0.199 to 0.529] | 0.202 [0.106 to 0.386]
Statistical Analysis 1: Comparison: Placebo vs Lanadelumab (DX-2930) 150 mg Every 4 Weeks; Test type: Other; p < 0.001, Chi-squared — p-values are adjusted for multiple testing; % change in mean rate (vs placebo) = -70.497, 95% CI 2-sided [-82.696 to -49.699] — % change in mean rate corresponds to 100% * (estimated mean rate ratio - 1); [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Lanadelumab (DX-2930) 300 mg Every 4 Weeks; Test type: Other; p < 0.001, Chi-squared — p-values are adjusted for multiple testing; % change in mean rate (vs placebo) = -73.285, 95% CI 2-sided [-84.316 to -54.496] — % change in mean rate corresponds to 100% * (estimated mean rate ratio - 1); [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Lanadelumab (DX-2930) 300 mg Every 2 Weeks; Test type: Other; p < 0.001, Chi-squared — p-values are adjusted for multiple testing; % change in mean rate (vs placebo) = -83.394, 95% CI 2-sided [-91.618 to -67.099] — % change in mean rate corresponds to 100% * (estimated mean rate ratio - 1); [other analysis details as in outcome 1, analysis 1]

4. Secondary Outcome: Rate of Investigator Confirmed Hereditary Angioedema (HAE) Attacks During Day 14 Through Day 182
Description: HAE attack was defined as a discrete episode during which the participant progressed from no angioedema to symptoms of angioedema. Rate of investigator confirmed HAE attacks during day 14 after study drug administration through day 182 was analyzed by the same poisson regression model as in the primary endpoint analysis.
Time Frame: From Day 14 to Day 182
Population: ITT population included all randomized participants who received any exposure to the investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: Attacks per 4 weeks
Arm/Group | Placebo | Lanadelumab (DX-2930) 150 mg Every 4 Weeks | Lanadelumab (DX-2930) 300 mg Every 4 Weeks | Lanadelumab (DX-2930) 300 mg Every 2 Weeks
Number analyzed (Participants) | 41 | 28 | 29 | 27
Attacks per 4 weeks | 1.988 [1.652 to 2.391] | 0.445 [0.283 to 0.698] | 0.489 [0.326 to 0.734] | 0.218 [0.115 to 0.414]
Statistical Analysis 1: Comparison: Placebo vs Lanadelumab (DX-2930) 150 mg Every 4 Weeks; Test type: Other; p < 0.001, Chi-squared — p-values are adjusted for multiple testing; % change in mean rate (vs placebo) = -77.622, 95% CI 2-sided [-86.253 to -63.572] — % change in mean rate corresponds to 100% * (estimated mean rate ratio - 1); [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Lanadelumab (DX-2930) 300 mg Every 4 Weeks; Test type: Other; p < 0.001, Chi-squared — p-values are adjusted for multiple testing; % change in mean rate (vs placebo) = -75.377, 95% CI 2-sided [-84.115 to -61.833] — % change in mean rate corresponds to 100% * (estimated mean rate ratio - 1); [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Lanadelumab (DX-2930) 300 mg Every 2 Weeks; Test type: Other; p < 0.001, Chi-squared — p-values are adjusted for multiple testing; % change in mean rate (vs placebo) = -89.008, 95% CI 2-sided [-94.325 to -78.707] — % change in mean rate corresponds to 100% * (estimated mean rate ratio - 1); [other analysis details as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to Day 182
Description: Adverse events were collected over the entire treatment period and were assigned to the treatment group without regard to the type of injection (that is placebo or active drug in the 150 mg q4wk and 300 mg q4wk groups). Number of adverse events were calculated as unique events per System Organ Class (SOC), preferred term (PT), participant and adverse event start date.
Arm/Group | Placebo | Lanadelumab (DX-2930) 150 mg Every 4 Weeks | Lanadelumab (DX-2930) 300 mg Every 4 Weeks | Lanadelumab (DX-2930) 300 mg Every 2 Weeks
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/28 | 0/29 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/41 | 0/28 | 3/29 | 2/27
Other Adverse Events (participants affected / at risk) | 40/41 | 25/28 | 26/29 | 23/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=41) | Lanadelumab (DX-2930) 150 mg Every 4 Weeks (N=28) | Lanadelumab (DX-2930) 300 mg Every 4 Weeks (N=29) | Lanadelumab (DX-2930) 300 mg Every 2 Weeks (N=27)
Hereditary angioedema (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bipolar ii disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=41) | Lanadelumab (DX-2930) 150 mg Every 4 Weeks (N=28) | Lanadelumab (DX-2930) 300 mg Every 4 Weeks (N=29) | Lanadelumab (DX-2930) 300 mg Every 2 Weeks (N=27)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (7) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (4) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Injection site bruising (General disorders) | 0 (0) | 3 (5) | 2 (2) | 1 (1)
Injection site discomfort (General disorders) | 0 (0) | 0 (0) | 2 (13) | 1 (10)
Injection site erythema (General disorders) | 1 (1) | 4 (23) | 2 (6) | 2 (7)
Injection site haematoma (General disorders) | 3 (3) | 1 (1) | 1 (2) | 1 (1)
Injection site haemorrhage (General disorders) | 1 (7) | 1 (2) | 0 (0) | 2 (11)
Injection site pain (General disorders) | 12 (71) | 13 (123) | 9 (68) | 14 (67)
Injection site paraesthesia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hereditary angioedema (Congenital, familial and genetic disorders) | 40 (577) | 17 (84) | 20 (108) | 15 (45)
Gastroenteritis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Otitis externa (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (3) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 11 (16) | 3 (5) | 7 (10) | 10 (12)
Procedural pain (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 3 (5) | 1 (1)
Headache (Nervous system disorders) | 8 (10) | 3 (10) | 5 (8) | 9 (18)
Migraine (Nervous system disorders) | 4 (4) | 2 (5) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (6):
  • Study Protocol: Original (2015-09-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT02586805/Prot_000.pdf
  • Study Protocol: Amendment 1 (2015-12-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT02586805/Prot_001.pdf
  • Study Protocol: Amendment 2 (2016-04-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT02586805/Prot_002.pdf
  • Study Protocol: Amendment 3 (2017-01-09): https://cdn.clinicaltrials.gov/large-docs/05/NCT02586805/Prot_003.pdf
  • Statistical Analysis Plan: Original (2016-05-24): https://cdn.clinicaltrials.gov/large-docs/05/NCT02586805/SAP_004.pdf
  • Statistical Analysis Plan: Amendment 1 (2017-05-03): https://cdn.clinicaltrials.gov/large-docs/05/NCT02586805/SAP_005.pdf